CLINICAL TRIAL: NCT01621139
Title: A Pilot Prospective Randomized Study to Evaluate the Effects of Acupuncture in Patients on Prolonged Mechanical Ventilation
Brief Title: A Pilot Clinical Trial to Evaluate the Effects of Acupuncture in Patients on Prolonged Mechanical Ventilation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-001937
Record Dates: First submitted 2012-03-29; First posted 2012-06-18 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Mechanical Ventilation Complication
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real acupuncture (Experimental): Real acupuncture group
  Interventions: Procedure: Acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture group
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Patients on mechanical ventilation greater than two days will be randomly assigned to real acupuncture group or sham acupuncture group

SUMMARY:
The purpose of this study is to investigate the role of acupuncture use on: 1) decrease the requirements for pharmacologic analgesic, 2) improve patient-reported pain, 3) expedite recovery process, and 4) improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

Consecutive male and post-menopausal female patients expected to require more than 24 hours of mechanical ventilation will be included.

Exclusion Criteria:

* Children < 18 years of age
* Patients with active resuscitation (fluid boluses greater than 2 Liter per hour, rapid transfusions, titration of vasoactive medication)
* Patients with hemodynamic instability: heart rate less than 40/min or greater than 120/min, SBP < 90 or > 180 mm Hg for longer than 2 continuous hours
* Patients who are pregnant or pre-menopausal
* Patients with expected survival less than 6 3 months
* Major deformities of the upper or lower extremities and/or any active skin lesions or ulcers in acupuncture treatment areas.
* Patients with a pacemaker or other implanted electronic device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
RASS (Richmond Agitation Sedation Scale) | baseline to six months

SECONDARY OUTCOMES:
ABPS (Aberdeen Back Pain Scale) | baseline to six months
Pain Scale | baseline to six months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States